CLINICAL TRIAL: NCT00980824
Title: ENGAGE - Meeting Mental Health Needs of Complex Comorbid Patients Attending A&E Following a Suicide Attempt. A Pilot Study.
Brief Title: ENGAGE - Meeting Mental Health Needs of Complex Comorbid Patients
Acronym: ENGAGE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: University of Glasgow, University of Glasgow
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 62060
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Comorbidity; Substance Abuse; Personality Disorder
Keywords: cognitive behaviour therapy; self harm; personality disorder; complex comorbidity; mental health
MeSH Terms: conditions — Substance-Related Disorders; Personality Disorders; Self-Injurious Behavior; Psychological Well-Being | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- therapy (Experimental): Cognitive behavioural therapy. Six sessions of structured focused therapy.
  Interventions: Behavioral: Cognitive behavioural therapy
- Standard treatment (Active Comparator): referral to specialised or generic mental health service
  Interventions: Other: Standard treatment

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy — Six sessions brief CBT.
  Arms: therapy
Other: Standard treatment — Referral to NHS services appropriate to patient's needs
  Arms: Standard treatment

SUMMARY:
Scotland has higher rates of suicide than other parts of the UK, an average rate of 15.1 per 100,000 in Scotland compared to 11.4 for England and Wales. The Scottish Government is committed to reducing suicide by 2013. Choose Life has led to staff in services such as Accident and Emergency (A&E) receiving recent training in suicide prevention through ASIST and STORM.

Evidence for interventions specific to A&E setting is limited despite the fact that this is the most likely point of first contact with health services for people at risk of this behaviour. Brief interventions that reduce repetition of self harm have not been particularly effective partly because of poor attendance and lack of focus on comorbidity. We propose to pilot an evaluation of a brief focused intervention, ENGAGE (based on MAnualised Cognitive Therapy,MACT, developed by the investigator (Kate Davidson) and Prof Ulrike Schmidt of the Institute of Psychiatry, London) for those who present at A&E with a suicide attempt and who have a complex presentation - a combination of substance abuse and or personality disorder, all of which are recognized as high risk factors for suicide. ENGAGE will specifically encourage patients to seek appropriate services to meet their mental health needs. This pilot will allow us to assess the feasibility of a full scale study.

DETAILED DESCRIPTION:
This is an exploratory single centre, randomised controlled trial of a complex intervention based on cognitive behavioural therapy principles for patients with a recent episode of suicide and who have personality disorder/s and or substance abuse (complex comorbidity). Patients who join the study will be randomly allocated to receive either ENGAGE CBT or Treatment as Usual (TAU). We will compare the effectiveness of ENGAGE with TAU. The primary outcome will be engagement with services - the number of contacts with mental health services (e.g. drug, alcohol and CMHT) in the 3 months following the participant's randomisation.

We will recruit 30 patients seen in the hospital by the Liaison Team with a suicide attempt who score above the threshold for personality disorder and drug or alcohol abuse using SAPAS,AUDIT and DAST assessments. If the patient is interested in the study a research assistant will obtain consent and conduct a baseline interview at which full personality disorder diagnostic status will be confirmed and further psychological measures will be taken. The patient will be randomised to ENGAGE (CBT) or TAU and interviewed again by the research assistant at 3 months post randomisation. The research assistant will be blind to treatment group. Those patients randomised to ENGAGE CBT will receive 6 sessions of the intervention from a CBT therapist. ENGAGE will help patients to identify problems, use problem solving to help prioritise and resolve problems and motivate patients to attend the treatment recommended by the liaison team. The ENGAGE therapist will encourage and, if necessary, facilitate patients with substance abuse and personality disorder to engage in the appropriate NHS services.

TAU - usual treatment is the services that patients may already be involved in or services that the patient has been referred to following the suicide episode.

ELIGIBILITY:
Inclusion Criteria:

* all patients will have had an episode of deliberate self harm
* test positive on either Drug Abuse Screening Test (DAST, Skinner 1982) or Alcohol Use Disorders Identification Test (AUDIT, Saunders 1983)

Exclusion Criteria:

* unable to give written informed consent
* unable to understand the purpose and nature of the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-09 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
The number of contacts with mental health services appropriate to the patient's needs. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kate M Davidson, PhD, Principal Investigator — University of Glasgow/NHS Greater Glasgow & Clyde
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, Lanarkshire, United Kingdom

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617